CLINICAL TRIAL: NCT03534869
Title: Auricular Acupuncture as Effective Pain Relief After Episiotomy: A Prospective Interventional Randomized Parallel Single-center Study
Brief Title: Auricular Acupuncture as Effective Pain Relief After Episiotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant in Otorhinolaryngology and Head and Neck Surgery, University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14280 / 16-4
Record Dates: First submitted 2018-04-30; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Acupuncture, Ear; Episiotomy; Complications; Pain, Labor
Keywords: auricular acupuncture; episiotomy; acupuncture; pain relief; analgesic therapy
MeSH Terms: conditions — Labor Pain | interventions — Acupuncture, Ear; Analgesics

STUDY DESIGN:
Intervention Model Description: The study was designed as a prospective interventional randomized parallel longitudinal single-center study to evaluate the effects of auricular acupuncture on pain relief after episiotomy conducted in the Department of Gynecology and Obstetrics, University Hospital Center Sestre milosrdnice, Zagreb, Croatia. Prospective data were collected from November 2016 to April 2017. The study included healthy pregnant women over 18 years of age, a minimum of 36 weeks gestation that underwent mediolateral episiotomy during vaginal delivery. Sixty patients were included in the study. The patients were allocated either of the groups by using a heads-tails binary result coin toss method. Twenty-nine patients were treated with auricular acupuncture for episiotomy pain relief combined with oral analgesic therapy per request, while 31 patients were treated with oral analgesics per request only. In both groups, administration of oral analgesics was recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ear Acupuncture and Oral Analgesics (Experimental): The acupuncture treatment consisted of three acupuncture needles on the dominant ear according to French auriculotherapy guidelines - internal genital area, external genital area and Shen Men point that is used to increase the anaesthetic effect according to both French and Chinese traditions.
  Additional oral analgesics (NSAID) could be supplied at any time upon patients request during hospitalization. Oral ibuprofen was given as first line therapy, while oral paracetamol was given as second line therapy.
  Interventions: Procedure: Ear acupuncture
- Oral Analgesics Only (Active Comparator): Postoperative standard oral analgesic therapy (NSAID) supplied at any time upon patients request during hospitalization. Oral ibuprofen would be given as first line therapy, while oral paracetamol would be given as second line therapy.
  Interventions: Drug: Analgesics

INTERVENTIONS:
Procedure: Ear acupuncture — French auriculotherapy guidelines - internal genital area, external genital area and Shen Men point.
  Other Names: Ear, acupuncture
  Arms: Ear Acupuncture and Oral Analgesics
Drug: Analgesics — Oral ibuprofen was given as first line therapy, while oral paracetamol was given as second line therapy.
  Other Names: Oral analgesics
  Arms: Oral Analgesics Only

SUMMARY:
Background: Episiotomy is performed in up to 30% of vaginal deliveries. Previously, pain treatment following episiotomy has relied on non-steroid anti-inflammatory drugs (NSAID) as analgesics, whose use during breastfeeding remains controversial due of their transfer to the child through lactation. The aim of the study is to determine the effect of acupuncture on postpartal perineal pain following episiotomy.

Methods: The study is designed as a prospective interventional randomized parallel single-center study to evaluate the effects of auricular acupuncture on pain relief after episiotomy. The population will encompass 60 patients that have had mediolateral episiotomy performed during vaginal delivery, with 29 receiving acupuncture therapy and 31 not receiving acupuncture therapy for pain relief. NSAID analgesic therapy will be made available per request.

DETAILED DESCRIPTION:
Study Protocol The study is designed as a prospective interventional randomized parallel longitudinal single-center study to evaluate the effects of auricular acupuncture on pain relief after episiotomy conducted in the Department of Gynecology and Obstetrics, University Hospital Center Sestre milosrdnice, Zagreb, Croatia. This institution performs up to 3100 deliveries per year. Episiotomy is indicated and performed in 30% of them.

Prospective data will be collected from November 2016 to April 2017. The study will include healthy pregnant women over 18 years of age, a minimum of 36 weeks' gestation that underwent mediolateral episiotomy during vaginal delivery. Sixty patients will be included in the study. Half of patients will be treated with auricular acupuncture for episiotomy pain relief and oral analgesics, while the other half will be treated with oral analgesics only. In both groups, administration of oral analgesics was recorded. The patients will be allocated to the groups by using a heads-tails coin toss.

In this study, auricular acupuncture will be used. The acupuncture treatment consists of three acupuncture needles on the dominant ear according to French auriculotherapy guidelines - internal genital area, external genital area and Shen Men point that is used to increase the anaesthetic effect according to both French and Chinese traditions (14,15). Acupuncture needles will be stimulated by manual rotation of the needle to evoke needle sensation De Qi. No electrostimulation will be used. Sterile 0,2 x 1,4 mm needles were used. The needles will be inserted within 6-8 hours after childbirth by a certified acupuncturist. The needles will be left in place until the hospital discharge of the patient on the third postpartal day, and removed by a certified acupuncturist.

Additional oral analgesics (NSAID) could be supplied at any time upon patients request during hospitalization. Oral ibuprofen would be given as first line therapy, while oral paracetamol would be given as second line therapy.

Primary outcome measures will be pain intensity (VAS score) immediately after birth, 2 hours after birth, during the first 3 days-at rest and activity. Secondary outcome measures will be the need for analgesics, the amount of given analgesics, and the number of analgesic repetitions during the day.

In addition, subjective experiences of postpartum bleeding and pain due to uterine contractions will be recorded. For those who had received acupuncture therapy, pain levels at the acupuncture site, analysis of acupuncture related experience included discomfort during sleep, other contacts with acupuncture previously and likelihood of recommending the method to a friend will be noted. After leaving the hospital, women in the acupuncture group will be asked to fill out a questionnaire on acupuncture treatment satisfaction. All patients will sign an informed consent form. Inter-group comparisons will be performed based on the patient status at the time of hospital admission and during hospital stay. Input parameters: age, education level, number of previous births. Characteristics of delivery will be noted as: the time of birth, the duration of the birth, the subjective experience of the birth, the application of epidural analgesia.

If labor starts before 8 AM, it will be considered as the first day of the hospitalization, and if labor starts later than 8 AM, the first day of hospitalization will be documented as the next day.

Pain intensity will be evaluated using the Visual Analog Scala score. VAS score is scaled from 1 (smallest pain) to 10 (strongest pain). VAS score higher than 3 was the cut-off point for analgesic administration. The patients will be divided into two groups based on their education level; the first group encompassing women who had finished high school, and the other women who hold a university degree.

Statistical analysis The results will be expressed as a number for categorical variables and as a median value (25th-75th interquartile range) for continuous variables. Continuous variables will be compared using the Student's t-test for independent samples, while categorical variables were compared using χ2-test. Fisher's exact test will be used if expected frequencies are less than five. All statistical tests will be two tailed, and P values < 0.05 considered statistically significant. All statistical analyses will be performed using MedCalc 9.5.1.0 (MedCalc Software, Mariakerke, Belgium).

Peer-reviewed publications containing data from the study have not yet been published.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women over 18 years of age
* a minimum of 36 weeks' gestation
* patients that underwent mediolateral episiotomy during vaginal delivery

Exclusion Criteria:

* any illness diagnosed during pregnancy
* unwillingness to submit to acupuncture therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy pregnant women over 18 years of age, a minimum of 36 weeks' gestation that underwent mediolateral episiotomy during vaginal delivery.
Enrollment: 60 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Pain relief | Immediately after birth, 2 hours after birth, during the first 3 days-at rest and activity.
  Level of pain intensity measured by VAS - Visual Analogue Scale score ranging from 1 (smallest pain level) to 10 (highest pain level).

SECONDARY OUTCOMES:
Oral analgesics amount | First 3 postpartal days.
  Amount of given analgesics in miligrams per patient per day during the first 3 postpartal days.
Postpartum bleeding and pain due to uterine contractions | First 3 postpartal days.
  Subjective levels of postpartum bleeding and pain due to uterine contractions recorded.
Number of analgesic repetitions during the day. | First 3 postpartal days.
  Number of times patients required oral analgesic therapy (N).

CONTACTS AND LOCATIONS:
Overall Officials: Andro Košec, MD, PhD, Study Chair — Department of Otorhinolaryngology and Head and Neck Surgery, University Hospital Center Sestre milosrdnice
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
All statistical data gathered from the study, no identifiable patient records.